CLINICAL TRIAL: NCT02478749
Title: Influence of Arm Retraction on the Relative Position of Clavicle and the Subclavian Vein,During Supraclavicular Approach for Central Venous Catheterization in Adults and Children
Brief Title: Influence of Arm Retraction on the Supraclavicular Approach for Subclavian Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H-1504-069-664
Record Dates: First submitted 2015-06-01; First posted 2015-06-23 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Subclavian Venous Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Infant (Experimental): patients aged younger than 1year
  Interventions: Procedure: arm retraction
- Child (Experimental): patients aged 1year to 5years
  Interventions: Procedure: arm retraction
- Adult (Experimental): adult patients
  Interventions: Procedure: arm retraction

INTERVENTIONS:
Procedure: arm retraction — gently pulling through the ipsilateral arm to the knee

SUMMARY:
The purpose of this study is to determine the effect of arm retraction on the supraclavicular approach for subclavian vein catheterization in adults and children.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia regardless of subclavian venous catheterization

Exclusion Criteria:

* patients with infection over the puncture site history of thoracic surgery or clavicular fracture vascular malformation anatomical abnormality of subclavian vein

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of distance between clavicle and confluence of internal jugular vein and subclavian vein while arm retraction | Outcome measure will be assessed during arm retraction and it would be within 30 second of arm retraction
Change in diameter of suvclavian vein at the confluence of internal jugular vein and subclavian vein | Outcome measure will be assessed during arm retraction and it would be within 30 second of arm retraction

CONTACTS AND LOCATIONS:
Overall Officials: Jintae Kim, MD.PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim EH, Lee JH, Song IK, Kim HC, Kim HS, Kim JT. Influence of caudal traction of ipsilateral arm on ultrasound image for supraclavicular central venous catheterization. Am J Emerg Med. 2016 May;34(5):851-5. doi: 10.1016/j.ajem.2016.01.038. Epub 2016 Feb 12. PMID 26947376